CLINICAL TRIAL: NCT06407154
Title: Chronical Illness-related Limitations of the Ability to Cope with Rising Temperatures: an Observational Study, Second Wave (CLIMATE-II)
Brief Title: Chronical Illness-related Limitations of the Ability to Cope with Rising Temperatures: an Observational Study, 2nd Wave
Acronym: CLIMATE-II
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: IPA-2024-01
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Coronary Disease; Myocardial Infarction; Heart Failure; Arrhythmias, Cardiac; Peripheral Artery Disease; Stroke; Ischemic Attack, Transient; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Pulmonary Disease, Chronic Obstructive; Asthma; Renal Insufficiency; Depressive Disorder; Anxiety Disorders; Schizophrenia; Peripheral Nervous System Diseases
MeSH Terms: conditions — Coronary Disease; Myocardial Infarction; Heart Failure; Arrhythmias, Cardiac; Peripheral Arterial Disease; Stroke; Ischemic Attack, Transient; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Pulmonary Disease, Chronic Obstructive; Asthma; Renal Insufficiency; Depressive Disorder; Anxiety Disorders; Schizophrenia; Peripheral Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The CLIMATE-II Observational Study examines to what extent chronically ill patients experience adverse health effects because of heat and whether the patients' specific health behavior, somatosensory amplification, risk and benefit perception, self-efficacy, health literacy, degree of urbanisation of the patients' administration district and characteristics of the patients' neighborhood are associated with these effects.

DETAILED DESCRIPTION:
The CLIMATE-II Observational Study aims to analyse to what extent chronically ill patients experience adverse health effects because of heat and whether the patients' specific health behavior, self-efficacy, or other factors are associated with these effects. This cohort study is based on an online survey of patients with chronic illness who are recruited in GP practices across all regions of Germany. After the baseline assessment, participants fill out symptom diaries on 12 specific days of observation over a maximum period of 12 weeks. The specific days of observation are selected based on the maximum temperature that can be expected within the respective weeks. The weather forecast will be checked every Thursday. If, in the upcoming 4 days, the maximum temperature is expected to exceed 30°C, the warmest day in this time frame will be chosen. Otherwise, the weather forecast will be checked again on Monday to choose the warmest of the remaining days of the week. On each day of observation, patients are notified by email at 6 pm.

Baseline assessment includes socio-demographic data, chronic diseases, health behavior, somatosensory amplification, perceived risk for adverse health effects because of heat, perceived benefit of protective behavior against heat, perceived social support, self-efficacy, and health literacy. Local data on temperatures and humidity will be assessed by the measurement stations of Germany's National Meteorological Service. Degree of urbanisation of administration districts is provided by the German Federal Institute for Research on Building, Urban Affairs and Spatial Development. Data will be analyzed by multivariable, multilevel regression analyses adjusted for possible confounders and random effects on the administration district and practice within administration district level.

ELIGIBILITY:
Inclusion Criteria:

* being 18 years or older
* at least one of the following conditions: Coronary Heart Disease; Myocardial Infarction; Heart Failure; Cardiac Arrhythmias; Peripheral Artery Disease; Stroke; Transient Ischemic Attack; Diabetes Mellitus (Type 1 or 2); Chronic Obstructive Pulmonary Disease; Asthma; Renal Insufficiency; Depressive Disorder; Anxiety Disorders; Schizophrenia; Peripheral Nervous System Diseases.

Exclusion Criteria:

* no capacity to consent
* severe visual impairment
* insufficient German language skills
* not able to use internet browser (eg, lack of hardware)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is located in different sites in Germany. Patients from approximately 80 GP practices will be included. In each practice, eligible patients receive a flyer including a QR-Code and a short link to register for the online study. After documenting informed consent within the application, patients fill out the baseline questionnaire and receive invitations for 12 subsequent assessments of symptoms by email. The investigators estimated that approximately 3,200 patients will be contacted. From experience with similar studies the investigators anticipated a response rate of 20% (=640 patients).
Sampling Method: Probability Sample
Enrollment: 578 (Actual)
Dates: Start 2024-05-21 (Actual); Primary Completion 2024-09-19 (Actual); Study Completion 2024-09-19 (Actual)

PRIMARY OUTCOMES:
Summary score of severity of adverse health effects | 15 May 2024 to 30 September 2024
  Observed adverse health effects include nausea, vomiting, tiredness/fatigue, vertigo, circulation problems/syncopes, muscle cramps, headache, extrasystoles, palpitations, edemas, shortness of breath, depressive mood, anxiety, and mental confusion. The severity in each symptom category is defined by the degree of limitations in usual activities from 0=none to 4=very severe. The summary score is calculated by adding the severity of each symptom category.

SECONDARY OUTCOMES:
Summary score of participants' implementation of protective behavior against heat | 15 May 2024 to 30 September 2024
  Implementation of protective behavior against heat is measured by agreement to nine statements, each rated from from 0=not at all to 3=completely. Statements include avoiding exposure to sun and heat (4 items), cooling strategies (2 items), clothing adjustment (1 item), avoiding physical exertion (1 item), and drinking enough (1 item). The summary score is calculated by adding the rating of all nine items.
Self-rated health | 15 May 2024 to 30 September 2024
  Subjective health condition on the day of assessment rated by participant on a visual analogue scale between 0 (worst possible) and 100 (best possible).
Level of medical service use | 15 May 2024 to 30 September 2024
  Level of service use is ordinally scaled and defined as 0=no service being used, 1=utilization of medical practices, 2=utilization of emergency departments, and 3=utilization of inpatient care. In case of multiple services being used, the highest category is chosen.
Number of participants who died | 15 May 2024 to 30 September 2024
  Participants are asked at baseline for permission to communicate with any confidential contact person in case they drop out from the study. Data about participants' death are derived from the contact persons' information about the reason for the participants' drop out of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Ingmar Schäfer, PD Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- Universitätsklinikum Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be available from the corresponding authors of study publications upon reasonable request.

REFERENCES:
- [Derived] Schafer I, Paucke V, Nothacker J, Menzel A, Dopfmer S, Hager K, Hueber S, Karimzadeh A, Kotter T, Loffler C, Muller BS, Scherer M, Luhmann D. Association between psychosocial factors and adverse effects of light-to-moderate ambient heat in patients with chronic diseases: results of the prospective cohort study CLIMATE-II. BMC Med. 2026 Jan 15. doi: 10.1186/s12916-026-04622-4. Online ahead of print. PMID 41540452